CLINICAL TRIAL: NCT00281359
Title: A Comparative Study of the Effectiveness of Treatment of Contractures With Mechanically Applied Stretch and Heat.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Action Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RL1 230
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; dynamic splinting; contractures; heat therapy
MeSH Terms: conditions — Cerebral Palsy; Contracture; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With heat (Experimental): heat applied to contracted tissues prior to using the active stretching orthosis.
  Interventions: Device: With heat
- Without heat (Placebo Comparator): No heat applied to the contracted tissues prior to using the stretching orthosis
  Interventions: Device: No heat

INTERVENTIONS:
Device: With heat — heat pad followed by dynamic splinting
  Other Names: heat pad followed by dynamic splinting
  Arms: With heat
Device: No heat — No heat added to tissue prior to dynamic splinting
  Arms: Without heat

SUMMARY:
This study is looking at new ways to stretch knee contractures in children with cerebral palsy using a specially designed splint.

DETAILED DESCRIPTION:
When using active orthoses to treat contractures, is the effectiveness of treatment improved by heating the contracted tissue prior to treatment?

ELIGIBILITY:
Inclusion Criteria:

children with cerebral palsy -

Exclusion Criteria:

absent thermal sensation -

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Range of motion | 12 weeks
  15 degree change in RoM

CONTACTS AND LOCATIONS:
Overall Officials: John Patrick, Principal Investigator — Robert Jones and Agnes Hunt Orthopaedic Hospital
Locations (1):
- Robert Jones and Agnes Hunt Orthopaedic and District Hospital NHS Trust, Oswestry, Shropshire, United Kingdom